CLINICAL TRIAL: NCT01884870
Title: The Impact of Silent Ureteral Stone on Renal Function and Kidney Anatomy: a Prospective Analysis
Brief Title: Silent Ureteral Stone: Impact on Renal Function and Kidney Anatomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Giovanni Scala Marchini, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 01187012.2.0000.0068; Online Number: 9015 (Registry Identifier: Online Number: 9015)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Urinary Calculi
Keywords: Asymptomatic; ureteral; calculi; renal function; treatment
MeSH Terms: conditions — Urinary Calculi; Calculi | interventions — Surgical Procedures, Operative; Endoscopy; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical Treatment (Other): Silent Ureteral Stone - Surgical Treatment
  Interventions: Procedure: Surgical Treatment

INTERVENTIONS:
Procedure: Surgical Treatment — Surgical Treatment - open, endoscopic or laparoscopic
  Other Names: Surgical Treatment - open, endoscopic or laparoscopic

SUMMARY:
Ureteral stones may be silent in 5.3% of patients. The goal of this study was to prospectively evaluate the impact of a silent ureteral stone on renal function.

DETAILED DESCRIPTION:
The prevalence of nephrolithiasis is increasing worldwide, reaching 5.2% in North America and 10.1% in Italy. The widespread use of computed tomography and ultrasonography have resulted in a greater detection rate of asymptomatic stones and, in part, might explain the trend. Clinically, kidney or ureteral stones range in severity from asymptomatic to presenting with complete renal failure. Therefore, it is not only the alarming incidence of urinary stone disease, but also the associated burden that makes this one of the most concerning conditions in public health.

The situation becomes even more distressing when managing asymptomatic stones. Studies of the natural history of stones have revealed that only 20% of patients yearly actually become symptomatic from a new stone, and one half of those require surgical intervention at some point. The guidelines are well established for the treatment of symptomatic urolithiasis, and many investigators have extensively studied the management of silent kidney stones. Conversely, the same is not true for silent ureterolithiasis. The purpose of the present study is to report the investigators experience managing silent ureteral stones and to prospectively analyze their true influence on renal function.

ELIGIBILITY:
Inclusion Criteria:

* Silent ureteral stone: no subjective/objective symptoms related to the ureteral calculi.
* Patient willing to participate in the study
* Complete pre/post-operative work-up

Exclusion Criteria:

* Treatment outside our institution
* No will to be a part of the study
* Incomplete pre/post-operative work-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral Renal Function | 1 year
  Ipsilateral renal function determined by dimercaptosuccinic acid scintigraphy (DMSA) 12 months after surgery.

SECONDARY OUTCOMES:
Serum Creatinine level | 1 year
  Serum Creatinine level
Estimated Creatinine Clearance | 1 year
  Estimated Creatinine Clearance
Renal Anatomy assessed by Ultrasound | 1 year
  Renal Anatomy assessed by Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni S Marchini, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinics Hospital - University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil